CLINICAL TRIAL: NCT05514119
Title: Fenofibrate to Prevent Ischemic Cholangiopathy in Donation After Circulatory Death Liver Transplantation (FICsDCD)
Brief Title: A Study to Assess the Role of Fenofibrate in Preventing Ischemic Cholangiopathy After Liver Transplantation
Acronym: FICsDCD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Channa R Jayasekera, MD, MSc, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-007122
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplant
Keywords: Ischemic Cholangiography
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recipients of DCD liver transplants (Experimental): Subjects that have undergone transplant of a liver donation after circulatory death (DCD) in the last 21-35 days will receive a 12 week fenofibrate (Lofibra) for a duration of 12 weeks
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — 160mg once daily orally for 12 weeks
  Other Names: Lofibra

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a once-daily medication, fenofibrate (Lofibra), to prevent ischemic cholangiography (IC) in persons who were transplanted with livers donated after circulatory death (DCD).

DETAILED DESCRIPTION:
In this prospective pilot study, we aim to evaluate 1) the tolerability and safety, 2) the efficacy of 12 weeks once-daily fenofibrate in reducing IC incidence after DCD liver transplantation, 3) assess the association between serum markers of cholestasis and development of IC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone Donation after Circulatory Death (DCD) liver transplantation (LT).
* At least one serum alkaline phosphatase level >2.5x upper limit of normal between post-LT days 21-60 (inclusive).

Exclusion criteria:

* LT performed for primary sclerosing cholangitis or primary biliary cholangitis.
* Untreated hepatic artery compromise (e.g thrombosis, stenosis)
* Untreated biliary anastomotic stricture or bile leak between days 0-60 after LT
* Renal dysfunction defined as baseline glomerular filtration rate < 30 ml/min.
* Previously known intolerance or allergy to fenofibrate.
* Other clinically significant comorbid condition, including psychiatric conditions, which in the opinion of the study team, may interfere with patient treatment, safety, assessment, or compliance with the treatment.
* Adults lacking capacity to consent to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Channa Jayasekera, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20537461

RESULTS

PARTICIPANT FLOW:
Groups:
- Recipients of DCD liver transplants: Subjects that underwent transplant of a liver donation after circulatory death (DCD) in the last 21-35 days received a 12 week fenofibrate (Lofibra) for a duration of 12 weeks
  Fenofibrate: 160mg once daily orally for 12 weeks
Period: Overall Study
Arm/Group | Recipients of DCD liver transplants
Started | 6
Completed | 5
Not Completed | 1
Not completed — Ineligible due to disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Recipients of DCD liver transplants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Fenofibrate
Description: Proportion of subjects to discontinue fenofibrate due to adverse events
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of DCD liver transplants
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Safety of Fenofibrate
Description: Proportion of subjects with a new grade 3 or 4 adverse event
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of DCD liver transplants
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Safety of Fenofibrate
Description: Proportion of subjects with acute cellular rejection during fenofibrate treatment
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of DCD liver transplants
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Safety of Fenofibrate
Description: Mean change in calculated glomerular filtration rate before, during and after fenofibrate treatment
Time Frame: Baseline, treatment weeks 4, 8, 12, and at 4 weeks after end of treatment
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Recipients of DCD liver transplants
Number analyzed (Participants) | 6
mL/min/1.73m^2
  Baseline | 75.3 (13.0)
  Treatment Week 4 | 62.7 (24.2)
  Treatment Week 8 | 62.2 (26.5)
  Treatment Week 12 | 51.4 (21.7)
  Post Treatment Week 4 | 60.5 (19.6)

5. Secondary Outcome: Safety of Fenofibrate
Description: Proportion of subjects myopathy confirmed by serum creatine kinase elevation
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients of DCD liver transplants
Number analyzed (Participants) | 6
Participants | 0

6. Secondary Outcome: Efficacy of Fenofibrate
Description: Incidence of ischemic cholangiopathy in those treated with 12 weeks of fenofibrate, compared to a historical control group
Time Frame: 12 weeks
Population: The historical cohort was not constructed due to inadequate enrollment of the treatment arm
Measure: Count of Participants; unit: Participants
Groups:
- Liver transplant recipients treated with fenofibrate: Subjects that underwent DCD liver transplantation in the preceding 21-35 days and were treated with 12 weeks of fenofibrate (Lofibra)
- Liver transplant patients not treated with fenofibrate (historical cohort): Subjects that underwent DCD liver transplantation between 1/1/2016-6/1/2021 and were not treated with fenofibrate
Arm/Group | Liver transplant recipients treated with fenofibrate | Liver transplant patients not treated with fenofibrate (historical cohort)
Number analyzed (Participants) | 6 | 0
Participants | 0 |

7. Secondary Outcome: The Number of Participants Who Developed Ischemic Cholangiopathy (IC)
Description: The number of participants who developed IC was assessed by measuring serum alkaline phosphatase, gamma glutamyl transferase, total bile acid level, fibroblast growth factor 19 level, and 7-alpha-hydroxy-cholesten-4 levels. Logistics regression was used to calculate the changes in serum alkaline phosphatase, gamma glutamyl transferase, total bile acid level, fibroblast growth factor 19 level, and 7-alpha-hydroxy-cholesten-4 and estimate the probability that a participant had developed IC. The probability can range from 0 (no development of IC) to 1 (development of IC), with a higher number indicating a worse outcome.
Time Frame: 12 weeks
Population: No participant developed ischemic cholangiopathy, precluding analysis
Measure: Count of Participants; unit: Participants
Groups:
- Alkaline phosphatase: Association between serum alkaline phosphatase level and development of ischemic cholangiopathy
- Serum gamma glutamyl transferase: Association between serum gamma glutamyl transferase level and development of ischemic cholangiopathy
- Total bile acid level: Association between total bile acid level and development of ischemic cholangiopathy
- Fibroblast growth factor-19 level: Association between fibroblast growth factor-19 level and development of ischemic cholangiopathy
- 7-alpha-hydroxy-cholesten-4 level: Association between 7-alpha-hydroxy-cholesten-4 level and development of ischemic cholangiopathy
Arm/Group | Alkaline phosphatase | Serum gamma glutamyl transferase | Total bile acid level | Fibroblast growth factor-19 level | 7-alpha-hydroxy-cholesten-4 level
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 16 weeks.
Arm/Group | Recipients of DCD liver transplants
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Study was terminated early due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT05514119/Prot_SAP_000.pdf